CLINICAL TRIAL: NCT04202211
Title: A Randomized Double-blind, Placebo-controlled Trial of Lyophilized Fecal Microbiota Transplantation for the Induction of Remission in Adults With Active Ulcerative Colitis
Brief Title: FMT for Remission of Active Ulcerative Colitis in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol changed substantially enough to warrant a separate submission
Sponsor: University of British Columbia (Other)
Collaborators: Crohn's and Colitis Canada (Other)
Responsible Party: Principal Investigator, Theodore Steiner, MD, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H19-03882
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: ulcerative colitis; Fecal Microbiota transplant; FMT; Inflammatory bowel disease; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo oral & enema (Placebo Comparator): twice weekly x 8 weeks: 10 placebo oral capsules + placebo enema
  Interventions: Other: Placebo oral; Other: Placebo enema
- LYO-FMT oral + placebo enema (Active Comparator): twice weekly x 8 weeks: 10 LYO-FMT oral capsules + 1 placebo enema
  Interventions: Biological: FMT oral; Other: Placebo enema
- LYO-FMT oral + LYO-FMT enema (Active Comparator): twice weekly x 8 weeks: 10 LYO-FMT oral capsules + 1 LYO-FMT enema
  Interventions: Biological: FMT oral; Biological: FMT enema

INTERVENTIONS:
Biological: FMT oral — lyophilized FMT given orally (10 capsules) twice weekly for total of 8 weeks
  Arms: LYO-FMT oral + LYO-FMT enema; LYO-FMT oral + placebo enema
Biological: FMT enema — lyophilized FMT given via enema (1) twice weekly for total of 8 weeks
  Arms: LYO-FMT oral + LYO-FMT enema
Other: Placebo oral — placebo given orally (10 capsules) twice weekly for total of 8 weeks
  Arms: Placebo oral & enema
Other: Placebo enema — placebo given via enema (1) twice weekly for total of 8 weeks
  Arms: LYO-FMT oral + placebo enema; Placebo oral & enema

SUMMARY:
The goal of this study is to establish the safety and effectiveness of lyophilized (LYO) fecal microbiota transplant (FMT) for treating ulcerative colitis (UC) in adults. The protocol is being re-designed to address relevant, current research questions in the context of FMT treatment for UC. Once a final protocol is approved, this webpage will be updated.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Willing and able to comply with all the required trial procedures
* Active ulcerative colitis as defined by Mayo score > 3 AND Mayo endoscopic sub-score > 1 (within 30 days before enrollment, or at baseline)

Exclusion Criteria:

* Planned or actively taking another investigational product
* Abdominal surgery within the past 60 days
* Patients with neutropenia with absolute neutrophil count <0.5 x 109/L at - Evidence of toxic megacolon or gastrointestinal perforation on imaging
* Peripheral white blood cell count > 35.0 x 109/L at enrollment AND temperature > 38.0oC
* Active infectious diarrhea at the time of enrolment
* Increase in medical therapy for UC within 3 months of enrollment. Continued treatment with stable dose of 5-ASA, azathioprine, 6-mercaptopurine, cyclosporine, prednisone and/or anti- TNF agents for at least 3 months of is allowed
* Severe UC requiring hospitalization at the time of enrolment
* Pregnant or lactating
* History of anaphylaxis to any food
* Requiring oral and/or intravenous systemic antibiotic therapy at the time of study enrolment
* Unwilling to discontinue probiotic (yogurt is allowed)
* Severe underlying disease such that the patient is not expected to survive for at least 30 days.
* Any condition that in the opinion of the investigator that would pose harm to the participant or the research staff for the potential participant to take part in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Remission of UC | 9 weeks following receipt of LYO-FMT
  achievement of remission of UC as defined by Mayo score ≤ 2 AND Mayo endoscopic score of ≤ 1

SECONDARY OUTCOMES:
Incidence/absence of adverse events upon treatment with LYO-FMT [safety and tolerability] | up to 5 years post-FMT
  Safety of LYO-FMT in patients with active UC as determined by absence of adverse events
UC disease progression | immediately after FMT (study) treatment period up to 5 years post-FMT
  Determine progression of UC based on development of any of the following:
  1. Clinical flare of UC requiring hospitalization up to 3 months post-FMT
  2. Increase in dosages of current UC specific medications up to 3 months' post FMT
  3. Time to colectomy for UC flare up to 12 months' post FMT
  4. Time to death directly attributable to UC up to 5 years post FMT
  5. Improvement in clinical response defined by decrease in Partial Mayo score by ≥ 3 points from pre to post LYO-FMT.
  6. Improvement in patient-reported health related QoL using Valuation of Lost Productivity and (VOLP) and RAND VR12 measured at pre and at 5 weeks, 12 and 24 weeks following LYO-FMT and annually for 5 years
  7. Reduction in biologic inflammatory markers (serum c-reactive protein (CRP) and fecal calprotectin) from pre to post LYO-FMT

CONTACTS AND LOCATIONS:
Overall Officials: Ted Steiner, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No